CLINICAL TRIAL: NCT01098045
Title: FDG/PET Imaging for the Assessment of Brown Adipose Tissue in HIV Lipodystrophy
Brief Title: HIV Fat Redistribution and the Evaluation of Brown Fat
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2009P-001836
Record Dates: First submitted 2010-03-25; First posted 2010-04-02 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: HIV Infections
Keywords: HIV; fat redistribution; brown adipose tissue; PET
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood tests will include a complete blood count, creatinine, SGPT TSH and Free T4, triglyceride, total, HDL and LDL cholesterol, HIV test, CD4 count (for HIV+ subjects only), HIV viral load (for HIV+ subjects only), fasting glucose, 2 hour OGTT, as well as tissue samples from fat biopsy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- HIV-infection with fat redistribution (lipoatrophy): 1. Evidence of HIV infection
  2. Age ≥ 20 and ≤ 60 years of age
  3. BMI measurement between 18-24 kg/m2
  4. HIV positive, on a stable HAART treatment regimen (including an NRTI) for > 12 months
  5. No evidence of fat redistribution rated by the investigator.
- Healthy controls: 1. No history of HIV infection
  2. Age ≥ 20 and ≤ 60 years of age
  3. BMI measurement between 18-29.9 kg/m2
- HIV-infected with fat redistribution (lipohypertrophy): 1. Evidence of HIV infection
  2. Age ≥ 20 and ≤ 60 years of age
  3. BMI measurement between 25-29.9 kg/m2
  4. HIV positive, on a stable HAART treatment regimen (including an NRTI) for > 12 months
  5. Evidence of significant fat redistribution rated by the investigator, including 1) significant fat atrophy of the face, arms or legs, and 2) significant increase in fat accumulation of the neck.
- Dicer Cohort: 30 men [HV-infected with fat redistribution (n = 10), HIV-infected without fat redistribution (n=10), and healthy controls (n= 10)] will be recruited for this group.

SUMMARY:
The specific aims of this study are to determine whether HIV-infected patients with significant fat redistribution and ectopic fat accumulation have increased brown adipose tissue using 18F-FDG Positron Emission Tomography techniques.

Recent studies suggest down regulation of Dicer, a major component of miRNA has an important role in the differentiation and function of brown and white adipose tissue and may contribute to lipodystrophy. Therefore we will expand on recent research in this area by recruiting HIV-infected men with lipodystrophy. We will perform subcutaneous fat biopsies of the dorsocervical and abdominal fat in a subset of HIV-infected and non-HIV-infected men in order to explore further the question of down regulation of Dicer and its implication on metabolic abnormalities in this population.

DETAILED DESCRIPTION:
Among individuals infected with HIV, highly active antiretroviral therapy has reduced the incidence of morbidity and mortality however, despite recent improvements in newer antiretrovirals patients continue to exhibit secondary effects related to body composition such as lipoatrophy of the periphery, increased adiposity of the trunk and lipomatosis, especially of the dorsocervical spine. Changes in body composition have been reported in 40-50% of HIV-infected patients. Several studies have shown that antiretroviral therapy contributes to changes in body composition and is coupled with increased dyslipidemia, insulin resistance and diabetes.

Accumulation of fat over the dorsocervical spine, or "buffalo" has been reported in 2% to 13% of HIV-infected patients. Enlargement of adipose tissue in the dorsocervical region involves subcutaneous fat and is therefore unique to fat accumulation of the abdominal area. Guallar et al. examined dorsocervical adipose tissue after surgical removal and found that adipose tissue in this area showed substantial levels of the marker gene of brown fat, uncoupling protein 1 (UCP-1) suggesting there may be brown adipose tissue (BAT) in HIV infected individuals with lipomatosis of the dorsocervical spine. Until recently, BAT was known to be present in rodents throughout their lifetime and was thought to be present in humans only during infancy and early childhood. However, recent studies using 18F-FDG PET-CT have confirmed the presence of BAT in adults. Brown adipose tissue is known to affect whole-body metabolism and may be related to insulin sensitivity as well as susceptibility to weight gain.

Using 18F-FDG PET techniques, our group has evaluated HIV-infected subjects with lipoatrophy and noted there was significantly increased glucose uptake into subcutaneous tissue which may suggest presence of BAT in HIV-infected patients. However our previous study did not specifically examine areas of BAT in the subjects. Therefore, using 18F-FDG PET-CT in addition to fat biopsies we propose to explore the presence of BAT in fat depots among HIV-infected patients with fat redistribution, focusing specifically in the cervical area.

Also, as recent studies suggest down regulation of Dicer, a major component of miRNA has an important role in the differentiation and function of brown and white adipose tissue and may contribute to lipodystrophy. We will perform subcutaneous fat biopsies of the dorsocervical and abdominal fat in a subset of HIV-infected and non-HIV-infected men in order to explore further the question of down regulation of Dicer and its implication on metabolic abnormalities in this population.

ELIGIBILITY:
Subject Selection and Enrollment:

Twenty male subjects comprised of four distinct groups will be recruited for the study. Subjects will be matched by age and body-mass index. The four groups are:

Group 1: HIV infected with fat redistribution (lipohypertrophy) (n=5) Group 2: HIV infected with fat redistribution (lipoatrophy) (n=5) Group 3: Healthy Controls (n=10)

Inclusion Criteria for HIV+ with fat redistribution (lipohypertrophy) subjects (Group 1)

1. Evidence of HIV infection
2. Age ≥ 20 and ≤ 60 years of age
3. BMI measurement between 25-29.9 kg/m2
4. HIV positive, on a stable HAART treatment regimen (including an NRTI) for > 12 months
5. Evidence of significant fat redistribution rated by the investigator, including 1) significant fat atrophy of the face, arms or legs, and 2) significant increase in fat accumulation of the neck.

Exclusion Criteria for HIV+ with fat redistribution (lipohypertrophy) (Group 1)

1. Hemoglobin < 10.0 g/dL
2. Diabetes or on medications for diabetes
3. Abnormal thyroid function
4. Therapy with medications such as beta blockers, alpha-blockers, sympatholytic drugs
5. Chronic adrenergic drug use (>3 months) and benzodiazepine use.
6. Therapy with glucocorticoids (oral and inhaled), growth hormone or other anabolic agents currently or within the past 3 months
7. Current substance abuse, including alcohol, cocaine and/or heroin
8. Other serious or chronic diseases
9. New antiretroviral regimen in the past 12 months
10. Any new serious opportunistic infection within the past 6 weeks

Inclusion Criteria for HIV+ with fat redistribution (lipoatrophy) (Group 2)

1. Evidence of HIV infection
2. Age ≥ 20 and ≤ 60 years of age
3. BMI measurement between 18-24 kg/m2
4. HIV positive, on a stable HAART treatment regimen (including an NRTI) for > 12 months
5. No evidence of fat redistribution rated by the investigator.

Exclusion Criteria for HIV+ with fat redistribution (lipoatrophy) (Group 2)

1. Hemoglobin < 10.0 g/dL
2. Diabetes or on medications for diabetes
3. Abnormal thyroid function
4. Therapy with medications such as beta blockers, alpha-blockers, sympatholytic drugs
5. Chronic adrenergic drug use (>3 months) and benzodiazepine use.
6. Therapy with glucocorticoids (oral and inhaled), growth hormone or other anabolic agents currently or within the past 3 months
7. Current substance abuse, including alcohol, cocaine and/or heroin
8. Other serious or chronic diseases
9. New antiretroviral regimen in the past 12 months
10. Any new serious opportunistic infection within the past 6 weeks

Inclusion Criteria for Healthy Controls (Group 3)

1. No history of HIV infection
2. Age ≥ 20 and ≤ 60 years of age
3. BMI measurement between 18-29.9 kg/m2

Exclusion Criteria for Healthy Controls (Group 3)

1. Hemoglobin <10.0 g/dL.
2. Diabetes or on medications for diabetes
3. Abnormal thyroid function.
4. Therapy with medications such as beta blockers, alpha-blockers, sympatholytic drugs
5. Chronic adrenergic drug use (>3 months) and benzodiazepine use.
6. Therapy with glucocorticoid (oral and inhaled), growth hormone or other anabolic agents currently or within the past 3 months
7. Current substance abuse, including alcohol, cocaine and/or heroin
8. Any history of serious or chronic diseases -

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: HIV infected patients with fat redistribution and non HIV controls
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-03; Primary Completion 2014-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Brown Fat | Baseline
  Brown Fat will be assessed by PET FDG

SECONDARY OUTCOMES:
UCP-1 | Baseline
  UCP-1 will be analyzed from tissue collected from a fat biopsy of dorsocervical spine fat accumulation.
Indirect Calorimetry | Baseline
  Indirect Calorimetry will be performed to measure resting energy expenditure
Anthropometrics | Baseline
  Anthropometric measurements of waist to hip ratio, leg circumference, arm circumference and neck circumference will be performed using a standardized technique.
Glucose tolerance | Baseline
  A baseline glucose level will be obtained and then patients will consume a 75g glucose beverage. Subjects must complete the beverage within 5-10 minutes. Subsequently, blood glucose at +30, +60, +90, and +120 minutes, insulin levels will be assessed at baseline and +120 minutes. Glucose tolerance will be calculated by insulin area under the curve in response to OGTT.
miRNAs | Baseline
  A baseline miRNA profile will be assessed and subsequent pathways

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital; Martin Torriani, MD, Study Director — Massachusetts General Hopsital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Mallon PW, Miller J, Cooper DA, Carr A. Prospective evaluation of the effects of antiretroviral therapy on body composition in HIV-1-infected men starting therapy. AIDS. 2003 May 2;17(7):971-9. doi: 10.1097/00002030-200305020-00005. PMID 12700446
- [Background] Bernasconi E, Boubaker K, Junghans C, Flepp M, Furrer HJ, Haensel A, Hirschel B, Boggian K, Chave JP, Opravil M, Weber R, Rickenbach M, Telenti A; Swiss HIV Cohort Study. Abnormalities of body fat distribution in HIV-infected persons treated with antiretroviral drugs: The Swiss HIV Cohort Study. J Acquir Immune Defic Syndr. 2002 Sep 1;31(1):50-5. doi: 10.1097/00126334-200209010-00007. PMID 12352150
- [Background] Lichtenstein KA, Ward DJ, Moorman AC, Delaney KM, Young B, Palella FJ Jr, Rhodes PH, Wood KC, Holmberg SD; HIV Outpatient Study Investigators. Clinical assessment of HIV-associated lipodystrophy in an ambulatory population. AIDS. 2001 Jul 27;15(11):1389-98. doi: 10.1097/00002030-200107270-00008. PMID 11504960
- [Background] Miller J, Carr A, Emery S, Law M, Mallal S, Baker D, Smith D, Kaldor J, Cooper DA. HIV lipodystrophy: prevalence, severity and correlates of risk in Australia. HIV Med. 2003 Jul;4(3):293-301. doi: 10.1046/j.1468-1293.2003.00159.x. PMID 12859330
- [Background] Friis-Moller N, Weber R, Reiss P, Thiebaut R, Kirk O, d'Arminio Monforte A, Pradier C, Morfeldt L, Mateu S, Law M, El-Sadr W, De Wit S, Sabin CA, Phillips AN, Lundgren JD; DAD study group. Cardiovascular disease risk factors in HIV patients--association with antiretroviral therapy. Results from the DAD study. AIDS. 2003 May 23;17(8):1179-93. doi: 10.1097/01.aids.0000060358.78202.c1. PMID 12819520
- [Background] Riddler SA, Smit E, Cole SR, Li R, Chmiel JS, Dobs A, Palella F, Visscher B, Evans R, Kingsley LA. Impact of HIV infection and HAART on serum lipids in men. JAMA. 2003 Jun 11;289(22):2978-82. doi: 10.1001/jama.289.22.2978. PMID 12799406
- [Background] Hadigan C, Meigs JB, Corcoran C, Rietschel P, Piecuch S, Basgoz N, Davis B, Sax P, Stanley T, Wilson PW, D'Agostino RB, Grinspoon S. Metabolic abnormalities and cardiovascular disease risk factors in adults with human immunodeficiency virus infection and lipodystrophy. Clin Infect Dis. 2001 Jan;32(1):130-9. doi: 10.1086/317541. Epub 2000 Dec 15. PMID 11118392
- [Derived] Srinivasa S, Torriani M, Fitch KV, Maehler P, Iyengar S, Feldpausch M, Cypess AM, Grinspoon SK. Brief Report: Adipogenic Expression of Brown Fat Genes in HIV and HIV-Related Parameters. J Acquir Immune Defic Syndr. 2019 Dec 15;82(5):491-495. doi: 10.1097/QAI.0000000000002180. PMID 31714428
- [Derived] Torriani M, Srinivasa S, Fitch KV, Thomou T, Wong K, Petrow E, Kahn CR, Cypess AM, Grinspoon SK. Dysfunctional Subcutaneous Fat With Reduced Dicer and Brown Adipose Tissue Gene Expression in HIV-Infected Patients. J Clin Endocrinol Metab. 2016 Mar;101(3):1225-34. doi: 10.1210/jc.2015-3993. Epub 2016 Jan 12. PMID 26756119
- [Derived] Torriani M, Zanni MV, Fitch K, Stavrou E, Bredella MA, Lim R, Cypess AM, Grinspoon S. Increased FDG uptake in association with reduced extremity fat in HIV patients. Antivir Ther. 2013;18(2):243-8. doi: 10.3851/IMP2420. Epub 2012 Oct 5. PMID 23041595